CLINICAL TRIAL: NCT02248662
Title: Impact of Radiation Therapy on Breast Conservation in DCIS
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Rinaa Punglia, MD MPH, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 12-420; CE-12-11-4173 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: DCIS
Keywords: DCIS; PCORI; ductal carcinoma in situ; radiation; oncology; patient-centered; decision aid; decision-making
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surveillance, Epidemiology, and End Results (SEER) Database: Data were obtained for women in Surveillance, Epidemiology, and End Results (SEER) with a diagnosis of ductal carcinoma in situ (DCIS) between 1990 and 2011 who had not undergone radiotherapy for DCIS and experienced a subsequent breast cancer or DCIS diagnosis.
- Surveillance, Epidemiology, and End Results (SEER)-Medicare: Data were obtained for women in Surveillance, Epidemiology, and End Results (SEER)-Medicare with a ductal carcinoma in situ (DCIS) diagnosis between 1991 and 2009 who had not undergone radiotherapy for DCIS and experienced a subsequent breast cancer or DCIS diagnosis.

SUMMARY:
Large regional variation exists in the use of radiotherapy after breast-conserving surgery (BCS) for ductal carcinoma in situ (DCIS). Although patients who do not receive initial radiotherapy for DCIS are candidates for subsequent BCS if they experience a second breast event, many undergo mastectomy instead.

DETAILED DESCRIPTION:
Patients and their physicians are often confronted with a decision between more intensive versus less intensive treatment for a particular diagnosis. Quality decision-making between these options requires careful balancing of the risks and side-effects, as well as weighing the expected outcomes and their associated value as assessed by the patient.

Although the incidence of DCIS has risen dramatically (1), there exists considerable debate about optimal treatment. In general, people with DCIS have high rates of recurrence-free survival. Intensive therapies for DCIS such as mastectomy (removal of the breast) or radiation therapy following BCS reduce the likelihood of a second breast diagnosis,(2-5) but have not been shown to improve survival.(6) In addition, radiation usually necessitates mastectomy should a new cancer or DCIS develop in the same breast at any point during the patient's lifetime. Patients also have a small chance of experiencing long-term toxicity. Previous radiation can also complicate reconstructive options following mastectomy. The tradeoff between risk of second breast diagnosis and side-effects and potential consequences of radiation therapy underscores the need for patient preference-driven decision making.

Patients who receive BCS alone without radiation therapy may be candidates for repeat BCS if they have a second breast event in the same breast. One study suggests that some women choose not to have radiation after DCIS because they want to preserve a breast-preservation option should a second breast diagnosis occur.(7) However, the likelihood of mastectomy versus BCS at time of new diagnosis in a previously un-irradiated breast is variable.(8-10) Whether a woman receives repeat breast-conserving surgery for a new diagnosis may not only be a function of the stage of diagnosis, but may be also determined by the regional treatment patterns used for management of DCIS. We sought to study whether regional intensity of radiation use for DCIS treatment increases the likelihood of mastectomy at time of second breast event, among women who have not received radiation therapy at initial DCIS diagnosis. (Punglia RS, Cronin AM, Uno H, et al. Association of Regional Intensity of Ductal Carcinoma In Situ Treatment With Likelihood of Breast Preservation. JAMA Oncol. Published online July 21, 2016.)

ELIGIBILITY:
This study used data from SEER and SEER-Medicare.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women identified from SEER and SEER-Medicare data with Stage 0-III breast cancer after DCIS who had received BCS without radiation for initial treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3436 (Actual)
Dates: Start 2013-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rinaa S. Punglia, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Harvard Pilgrim Health Care Institute, Boston, Massachusetts
  - Dartmouth College, Hanover, New Hampshire
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sumner WE 3rd, Koniaris LG, Snell SE, Spector S, Powell J, Avisar E, Moffat F, Livingstone AS, Franceschi D. Results of 23,810 cases of ductal carcinoma-in-situ. Ann Surg Oncol. 2007 May;14(5):1638-43. doi: 10.1245/s10434-006-9316-1. Epub 2007 Jan 24. PMID 17245612
- [Background] Kim SY, Han BK, Kim EK, Choi WJ, Choi Y, Kim HH, Moon WK. Breast Cancer Detected at Screening US: Survival Rates and Clinical-Pathologic and Imaging Factors Associated with Recurrence. Radiology. 2017 Aug;284(2):354-364. doi: 10.1148/radiol.2017162348. Epub 2017 Apr 6. PMID 28387638
- [Background] EORTC Breast Cancer Cooperative Group; EORTC Radiotherapy Group; Bijker N, Meijnen P, Peterse JL, Bogaerts J, Van Hoorebeeck I, Julien JP, Gennaro M, Rouanet P, Avril A, Fentiman IS, Bartelink H, Rutgers EJ. Breast-conserving treatment with or without radiotherapy in ductal carcinoma-in-situ: ten-year results of European Organisation for Research and Treatment of Cancer randomized phase III trial 10853--a study by the EORTC Breast Cancer Cooperative Group and EORTC Radiotherapy Group. J Clin Oncol. 2006 Jul 20;24(21):3381-7. doi: 10.1200/JCO.2006.06.1366. Epub 2006 Jun 26. PMID 16801628
- [Background] Fisher B, Land S, Mamounas E, Dignam J, Fisher ER, Wolmark N. Prevention of invasive breast cancer in women with ductal carcinoma in situ: an update of the National Surgical Adjuvant Breast and Bowel Project experience. Semin Oncol. 2001 Aug;28(4):400-18. doi: 10.1016/s0093-7754(01)90133-2. PMID 11498833
- [Background] Emdin SO, Granstrand B, Ringberg A, Sandelin K, Arnesson LG, Nordgren H, Anderson H, Garmo H, Holmberg L, Wallgren A; Swedish Breast Cancer Group. SweDCIS: Radiotherapy after sector resection for ductal carcinoma in situ of the breast. Results of a randomised trial in a population offered mammography screening. Acta Oncol. 2006;45(5):536-43. doi: 10.1080/02841860600681569. PMID 16864166
- [Background] Houghton J, George WD, Cuzick J, Duggan C, Fentiman IS, Spittle M; UK Coordinating Committee on Cancer Research; Ductal Carcinoma in situ Working Party; DCIS trialists in the UK, Australia, and New Zealand. Radiotherapy and tamoxifen in women with completely excised ductal carcinoma in situ of the breast in the UK, Australia, and New Zealand: randomised controlled trial. Lancet. 2003 Jul 12;362(9378):95-102. doi: 10.1016/s0140-6736(03)13859-7. PMID 12867108
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Correa C, McGale P, Taylor C, Wang Y, Clarke M, Davies C, Peto R, Bijker N, Solin L, Darby S. Overview of the randomized trials of radiotherapy in ductal carcinoma in situ of the breast. J Natl Cancer Inst Monogr. 2010;2010(41):162-77. doi: 10.1093/jncimonographs/lgq039. PMID 20956824
- [Background] Kaplan CP, Napoles AM, Hwang ES, Bloom J, Stewart S, Nickleach D, Karliner L. Selection of treatment among Latina and non-Latina white women with ductal carcinoma in situ. J Womens Health (Larchmt). 2011 Feb;20(2):215-23. doi: 10.1089/jwh.2010.1986. Epub 2010 Dec 3. PMID 21128819
- [Background] Fisher B, Dignam J, Wolmark N, Mamounas E, Costantino J, Poller W, Fisher ER, Wickerham DL, Deutsch M, Margolese R, Dimitrov N, Kavanah M. Lumpectomy and radiation therapy for the treatment of intraductal breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-17. J Clin Oncol. 1998 Feb;16(2):441-52. doi: 10.1200/JCO.1998.16.2.441. PMID 9469327
- [Background] Fong J, Kurniawan ED, Rose AK, Mou A, Collins JP, Miller JA, Mann GB. Outcomes of screening-detected ductal carcinoma in situ treated with wide excision alone. Ann Surg Oncol. 2011 Dec;18(13):3778-84. doi: 10.1245/s10434-011-1748-6. Epub 2011 Jun 1. PMID 21630124
- [Background] Wong JS, Kaelin CM, Troyan SL, Gadd MA, Gelman R, Lester SC, Schnitt SJ, Sgroi DC, Silver BJ, Harris JR, Smith BL. Prospective study of wide excision alone for ductal carcinoma in situ of the breast. J Clin Oncol. 2006 Mar 1;24(7):1031-6. doi: 10.1200/JCO.2005.02.9975. Epub 2006 Feb 6. PMID 16461781
- [Background] Pickle LW, MungioleM, Jones GK, White AA. Atlas of United States Mortality. Hyattsville, MD: Centers for Disease Control and Prevention; December 1996. http://www.cdc.gov/nchs/data/misc/atlasmet.pdf. Accessed September 1, 2015.
- [Background] Wennberg JE, Fisher ES, Skinner JS. Geography and the debate over Medicare reform. Health Aff (Millwood). 2002 Jul-Dec;Suppl Web Exclusives:W96-114. doi: 10.1377/hlthaff.w2.96. PMID 12703563
- [Background] Jagsi R, Abrahamse P, Hawley ST, Graff JJ, Hamilton AS, Katz SJ. Underascertainment of radiotherapy receipt in Surveillance, Epidemiology, and End Results registry data. Cancer. 2012 Jan 15;118(2):333-41. doi: 10.1002/cncr.26295. Epub 2011 Jun 29. PMID 21717446

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The computer model included data from sources including the NSABP B-17 and B-24 trials; the UK, Australia, and New Zealand ductal carcinoma in situ (DCIS) trial; an observational study of newly diagnosed patients with DCIS treated in British Columbia; and SEER databases. The researchers also conducted two retrospective studies.
Pre-assignment Details: Originally, 38,514 total records from each database used for this study were screened for enrollment into the final cohort. After eligibility criteria were applied to the sample, the final sample size was 3,436.
Groups:
- Surveillance Epidemiology and End Results (SEER)-Medicare: SEER-Medicare diagnoses from 1990-2009 linked to Medicare claims through 2010
  Breast Conserving Surgery +/- Radiotherapy or Mastectomy for secondary breast cancer
- Surveillance Epidemiology and End Results (SEER): Data was collected from the Surveillance Epidemiology and End Results (SEER) database on patients with ductal carcinoma in situ (DCIS) between 1990 and 2011.
  Breast Conserving Surgery +/- Radiotherapy or Mastectomy for secondary breast cancer
Period: Overall Study
Arm/Group | Surveillance Epidemiology and End Results (SEER)-Medicare | Surveillance Epidemiology and End Results (SEER)
Started | 5320 | 33194
Completed | 757 | 2679
Not Completed | 4563 | 30515

BASELINE CHARACTERISTICS:
Groups:
- SEER: Data was collected from the Surveillance Epidemiology and End Results database on patients with DCIS between 1990 and 2011.
- SEER-Medicare: SEER-Medicaid diagnoses from 1990-2009 linked to Medicare claims through 2010
- Total: Total of all reporting groups
Arm/Group | SEER | SEER-Medicare | Total
Number analyzed (Participants) | 2679 | 757 | 3436
Age, Customized [Count of Participants; unit: Participants]
  Age at Secondary Diagnosis: <50 years | 363 | 0 | 363
  Age at Secondary Diagnosis: 50 to 59 years | 605 | 0 | 605
  Age at Secondary Diagnosis: 60 to 69 years | 679 | 63 | 742
  Age at Secondary Diagnosis: 70 to 90 years | 1032 | 694 | 1726
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2679 | 757 | 3436
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 216 | 42 | 258
  Not Hispanic or Latino | 2463 | 715 | 3178
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 2133 | 658 | 2791
  Race: Black | 283 | 64 | 347
  Race: Other | 263 | 35 | 298
Number of Participants with Household Income Within Census Data Quintiles [Count of Participants; unit: Participants] — Participants' median income levels were assessed using US Census Data. Income data was gathered from census tract information. The census tract data was then put into quintiles ranging from lowest socioeconomic status (quintile 1) to highest socioeconomic status (quintile 5).
  Participants
    1 (lowest) | 763 | 137 | 900
    2 | 301 | 157 | 458
    3 | 461 | 153 | 614
    4 | 608 | 133 | 741
    5 (highest) | 546 | 177 | 723
Number of Participants in Education Levels Within Census Data Quintiles [Count of Participants; unit: Participants] — Participants' education levels were assessed using US Census Data. Education data was gathered from census tract information. The census tract data was then put into quintiles ranging from lowest education level (quintile 1) to highest education level (quintile 5).
  Participants
    1 (lowest) | 664 | 156 | 820
    2 | 490 | 167 | 657
    3 | 459 | 143 | 602
    4 | 514 | 148 | 662
    5 (highest) | 552 | 143 | 695
Residence [Count of Participants; unit: Participants]
  Urban | 2560 | 701 | 3261
  Rural | 119 | 56 | 175
Number of Participants with a Secondary SEER Diagnosis [Count of Participants; unit: Participants]
  No | 0 | 370 | 370
  Yes | 2679 | 387 | 3066
Number of Participants with Secondary SEER Diagnoses and Staging [Count of Participants; unit: Participants] — For the SEER-Medicare sample, frequencies and percentages are calculated only among patients with a secondary SEER diagnosis. The number of cases who had a secondary SEER diagnosis was less than the number of cases included in this cohort at baseline. Sometimes, it was clear that patients had a secondary SEER diagnosis, but the stage was unclear. The total number of SEER-Medicare cases in the final analysis was 387. Staging in the SEER and SEER-Medicare data registries is consistent with general cancer staging. Higher stages indicate worse outcomes. Population: The number of cases with a secondary SEER diagnosis was less than the number of cases included in this cohort at baseline. Sometimes, it was clear that patients had a secondary SEER diagnosis, but the stage was unclear. The total number of SEER-Medicare cases in the final analysis was 387.
  Participants
    Ductal carcinoma in situ (DCIS): number analyzed (Participants) | 2679 | 387 | 3066
    Ductal carcinoma in situ (DCIS) | 843 | 111 | 954
    Stage I: number analyzed (Participants) | 2679 | 387 | 3066
    Stage I | 1185 | 177 | 1362
    Stage II-III: number analyzed (Participants) | 2679 | 387 | 3066
    Stage II-III | 523 | 71 | 594
    Unknown: number analyzed (Participants) | 2679 | 387 | 3066
    Unknown | 128 | 28 | 156
Number of Participants with ER Status for Secondary SEER Diagnosis [Count of Participants; unit: Participants] — For the SEER-Medicare sample, frequencies and percentages are calculated only among patients with a secondary SEER diagnosis. The total number of cases who had ER status information was less than the overall number of cases included in this cohort at baseline. Analysis was performed only on the number of cases that had a secondary SEER diagnosis. In some instances, it was clear patients had a secondary SEER diagnosis, but it was not clear whether the diagnosis was ER positive or negative. Therefore, the total number of SEER-Medicare cases in the final analysis was 387. Population: The total number of cases with ER status information was less than the overall number of cases included in this cohort at baseline. Analysis was performed only on the number of cases that had a secondary SEER diagnosis. In some instances, it was clear patients had a secondary SEER diagnosis, but it was unclear whether the diagnosis was ER+ or ER-.
  Participants
    Positive: number analyzed (Participants) | 2679 | 387 | 3066
    Positive | 1675 | 227 | 1902
    Negative: number analyzed (Participants) | 2679 | 387 | 3066
    Negative | 324 | 42 | 366
    Unknown: number analyzed (Participants) | 2679 | 387 | 3066
    Unknown | 680 | 118 | 798
Number of Participants with Laterality for Secondary SEER Diagnosis [Count of Participants; unit: Participants] — For the SEER-Medicare sample, frequencies and percentages are calculated only among patients with laterality information. The total number of cases who had laterality information was less than the number of cases included in this cohort. Analysis was performed only on the number of cases that had a secondary SEER diagnosis. In some instances, it was clear patients had a secondary SEER diagnosis, but it was not clear whether the diagnosis was ipsilateral or contralateral. Therefore, the total number of SEER-Medicare cases in the final analysis was 387. Population: The total number of cases with laterality information was less than the number of cases included in this cohort. Analysis was performed only on the number of cases that had a secondary SEER diagnosis. In some instances, it was clear patients had a secondary SEER diagnosis, but it was not clear whether the diagnosis was ipsilateral or contralateral.
  Participants
    Ipsilateral: number analyzed (Participants) | 2679 | 387 | 3066
    Ipsilateral | 1619 | 239 | 1858
    Contralateral: number analyzed (Participants) | 2679 | 387 | 3066
    Contralateral | 1060 | 148 | 1208
Year of secondary diagnosis [Count of Participants; unit: Participants]
  1990-1995 | 133 | 47 | 180
  1996-2000 | 426 | 128 | 554
  2001-2005 | 778 | 263 | 1041
  2006-2011 | 1342 | 319 | 1661
Interval between diagnoses [Mean (Inter-Quartile Range); unit: years] | 4.6 [2.3 to 7.6] | 2.4 [1.1 to 4.6] | NA [NA to NA] — This data was not calculated and was not included in the final, published article. The raw data was from SEER, and is no longer available to calculate this value because our data usage agreement with SEER expired.
Treatment intensity for primary DCIS [Count of Participants; unit: Participants] — Regional treatment intensity was measured by using health service areas (HSAs). HSAs were assiged to 1 of 3 clusters based on the observed proportion of radiotherapy used as coded by SEER and SEER-Medicare. The HSAs with the highest proportion of patients receiving radiotherapy were assigned to the high cluster; those with the lowest to the low cluster. This table shows how many people lived in each HSA.
  Participants
    Low (HSAs with lowest proportion receiving RT) | 966 | 261 | 1227
    Medium | 885 | 274 | 1159
    High (HSAs with highest proportion receiving RT) | 828 | 222 | 1050
Charlson comorbidity score [Count of Participants; unit: Participants] — The Charlson comorbidity score is used to predict the risk of death within 1 year of hospitalization for patients with specific comorbid conditions. A high score indicates increased risk. Population: Data was not collected for the SEER group and the data is no longer available to us.
  Participants
    0-1: number analyzed (Participants) | 0 | 757 | 757
    0-1 |  | 686 | 686
    2+: number analyzed (Participants) | 0 | 757 | 757
    2+ |  | 71 | 71
Distance to nearest radiation facility [Count of Participants; unit: Participants] — Population: Data was not collected for the SEER group and is no longer available to us.
  Participants
    <10 miles: number analyzed (Participants) | 0 | 757 | 757
    <10 miles |  | 634 | 634
    10+ miles: number analyzed (Participants) | 0 | 757 | 757
    10+ miles |  | 123 | 123
Chemotherapy for secondary breast event [Count of Participants; unit: Participants] — Population: Data was not collected for the SEER group and the data is no longer available to us.
  Participants
    No: number analyzed (Participants) | 0 | 757 | 757
    No |  | 719 | 719
    Yes: number analyzed (Participants) | 0 | 757 | 757
    Yes |  | 38 | 38
MRI in 6 months before secondary breast event [Count of Participants; unit: Participants] — Population: Data was not collected for the SEER group and the data is no longer available to us.
  Participants
    No: number analyzed (Participants) | 0 | 757 | 757
    No |  | 706 | 706
    Yes: number analyzed (Participants) | 0 | 757 | 757
    Yes |  | 51 | 51

OUTCOME MEASURES:

1. Primary Outcome: Association Between Patient Characteristics and Three-Level Cluster of Treatment Intensity for Primary DCIS
Description: The investigators defined treatment intensity in a health services area to be the proportion of patients undergoing breast conserving surgery for DCIS who receive radiation therapy. Because a proportion is challenging to analyze statistically given that the precision of the estimate depends on the size of the denominator which varies across service areas, we used hierarchical modeling to categorize the health service areas into three categories (low, medium, high), using a latent variable to determine which health service area belongs to each of the three categories. The cutoffs separating the groups were based on the hierarchical model, taking the precision of the estimated proportion of patients receiving radiation into account. Health service areas with the highest proportions of patients receiving radiation were assigned to the "high" cluster; those with the lowest proportions to the "low" cluster; and those in the between to the "medium" cluster.
Time Frame: 20 Years
Measure: Count of Participants; unit: Participants
Groups:
- SEER - Low Treatment Cluster; SEER-Medicare - Low Treatment Cluster: Low treatment intensity for primary DCIS
- SEER-Medium Treatment Cluster; SEER-Medicare - Medium Treatment Cluster: Medium treatment intensity for primary DCIS
- SEER - High Treatment Cluster; SEER Medicare - High Treatment Cluster: High treatment intensity for primary DCIS
Arm/Group | SEER - Low Treatment Cluster | SEER-Medium Treatment Cluster | SEER - High Treatment Cluster | SEER-Medicare - Low Treatment Cluster | SEER-Medicare - Medium Treatment Cluster | SEER Medicare - High Treatment Cluster
Number analyzed (Participants) | 966 | 885 | 828 | 222 | 274 | 261
Participants
  Age at secondary diagnosis: <50 | 145 | 115 | 99 | 0 | 0 | 0
  Age at secondary diagnosis:50 to 59 | 213 | 230 | 157 | 0 | 0 | 0
  Age at secondary diagnosis: 60 to 69 | 232 | 221 | 232 | 11 | 19 | 31
  Age at secondary diagnosis: 70 to 90 | 377 | 318 | 339 | 211 | 255 | 230
  Race: White | 715 | 752 | 662 | 191 | 252 | 217
  Race: Black | 106 | 71 | 99 | 16 | 16 | 34
  Race: Other | 135 | 62 | 66 | 16 | 8 | 13
  Hispanic: No | 831 | 823 | 811 | 206 | 258 | 251
  Hispanic: Yes | 135 | 62 | 17 | 16 | 16 | 10
  Median income: Quintile 1 (lowest) | 570 | 80 | 108 | 31 | 36 | 68
  Median income: Quintile 2 | 10 | 97 | 190 | 33 | 71 | 52
  Median income: Quintile 3 | 39 | 212 | 215 | 42 | 63 | 47
  Median income: Quintile 4 | 222 | 221 | 157 | 40 | 52 | 42
  Median income: Quintile 5 (highest) | 116 | 274 | 157 | 73 | 55 | 50
  High school educated, Quintile 1 (lowest) | 551 | 62 | 58 | 31 | 36 | 68
  High school educated, Quintile 2 | 222 | 106 | 157 | 33 | 71 | 55
  High school educated, Quintile 3 | 39 | 212 | 215 | 42 | 63 | 47
  High school educated, Quintile 4 | 10 | 319 | 132 | 40 | 52 | 48
  High school educated, Quintile 5 (highest) | 116 | 274 | 157 | 73 | 55 | 50
  Residence: Urban | 947 | 858 | 762 | 218 | 258 | 224
  Residence: Rural | 19 | 27 | 66 | 4 | 16 | 37
  Secondary SEER Diagnosis: No | 0 | 0 | 0 | 98 | 132 | 141
  Secondary SEER Diagnosis: Yes | 966 | 885 | 828 | 124 | 142 | 120
  Stage of secondary SEER Diagnosis: DCIS | 290 | 274 | 282 | 31 | 47 | 34
  Stage of secondary SEER Diagnosis: Stage I | 425 | 395 | 364 | 60 | 63 | 55
  Stage of secondary SEER Diagnosis: Stage II-III | 213 | 177 | 132 | 24 | 22 | 23
  Stage of secondary SEER Diagnosis: Unknown | 48 | 35 | 50 | 9 | 11 | 8
  ER status of secondary SEER diagnosis: Positive | 609 | 566 | 497 | 75 | 85 | 68
  ER status of secondary SEER diagnosis: Negative | 106 | 124 | 99 | 11 | 14 | 16
  ER status of secondary SEER diagnosis: Unknown | 251 | 195 | 232 | 38 | 44 | 37
  Laterality of secondary SEER diagnosis:Ipsilateral | 580 | 522 | 513 | 82 | 88 | 70
  Laterality of secondary SEER diag.: Contralateral | 386 | 363 | 315 | 42 | 55 | 50
  Year of secondary diag.: 1990-1995 | 39 | 35 | 58 | 20 | 11 | 16
  Year of secondary diag.: 1996-2000 | 145 | 97 | 190 | 31 | 52 | 44
  Year of secondary diag.: 2001-2005 | 319 | 239 | 215 | 82 | 88 | 91
  Year of secondary diag.: 2006-2011 | 464 | 513 | 364 | 89 | 121 | 110
  Charlson comorbidity score: 0-1 | 0 | 0 | 0 | 202 | 252 | 232
  Charlson comorbidity score: 2+ | 0 | 0 | 0 | 20 | 22 | 29
  Distance to nearest radiation facility: <10 mi | 0 | 0 | 0 | 206 | 225 | 201
  Distance to nearest radiation facility: 10+ mi | 0 | 0 | 0 | 16 | 49 | 60
  Chemotherapy for secondary breast event: No | 0 | 0 | 0 | 209 | 260 | 251
  Chemotherapy for secondary breast event: Yes | 0 | 0 | 0 | 18 | 16 | 18
Statistical Analysis 1: Comparison: SEER - Low Treatment Cluster vs SEER-Medicare - Low Treatment Cluster; Unadjusted associations between patient characteristics and the three-level cluster of treatment intensity for primary DCIS were evaluated using Chi-squared tests. We used multivariable modeling to adjust for potential confounders. We also conducted a sensitivity analysis using propensity score matching to balance regional treatment intensity for primary DCIS with respect to the covariates included in the multivariable models; Test type: Other — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; p < 0.05, Regression, Logistic — A two-sided p value of less than 0.05 was considered to indicate statistical significance; Adjusted percentages for receipt of mastectomy were calculated by setting covariates to their observed mean values; Odds Ratio (OR) = 1.00 — This group is the reference group
Statistical Analysis 2: Comparison: SEER-Medium Treatment Cluster vs SEER-Medicare - Medium Treatment Cluster; [analysis description as in outcome 1, analysis 1]; Test type: Other — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; p < 0.05, Chi-squared — A two-sided p value of less than 0.05 was considered to indicate statistical significance; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.71 to 1.56]
Statistical Analysis 3: Comparison: SEER - High Treatment Cluster vs SEER Medicare - High Treatment Cluster; Test type: Other; p < 0.05, Chi-squared; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.27 to 2.84]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: This was a retrospective review of data from the SEER and SEER-Medicare registries. There were no adverse events to report because this was not a clinical trial.
Groups:
- SEER; SEER-Medicare: Breast conservation surgery +/- Radiotherapy or Mastectomy for secondary breast cancer
Arm/Group | SEER | SEER-Medicare
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No data set can capture all of the complexity surrounding surgical decision making at the time of a second diagnosis. We did not have information about patient preferences or the clinical characteristics about second breast event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No